CLINICAL TRIAL: NCT02366650
Title: Help in the Emergency Room to Detect Organ Dysfunction - The HERO Study
Brief Title: Help in the Emergency Room to Detect Organ Dysfunction
Acronym: HERO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Adam Linder, MD,PhD, Region Skane
Other Study IDs: HERO1
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Sepsis; Critical Illness
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lund ED: appr 100-200 patients at Lund ED
- Helsingborg ED: appr 100-200 patients at Helsingborg ED
- Vancouver ED: appr 100 patients at St Paul's hospital ED
- Bern ED: appr 100 patients at Bern ED

SUMMARY:
The purpose of this prospective, non-interventional clinical study is to assess the clinical validity of a number of markers (including Heparin Binding Protein (HBP), Procalcitonin (PCT), C-reactive protein (CRP), White cell count (WCC) and lactate) for indicating the presence of organ dysfunction, or outcome, of patients with organ dysfunctions following emergency department admission or hospitalization. Secondary objectives are to identify novel putative biomarkers and to identify risk factors for negative long-term effects of acute critical illness The HBP assay is an enzyme-linked immunosorbent assay (ELISA) for the quantitative determination of Heparin Binding Protein in human plasma.

ELIGIBILITY:
Inclusion Criteria:

i) ≥18 years of age ii) 1 or more of the following criteria: Saturation<90% without oxygen or <93% with oxygen or reported saturation<90%, Respiratory frequency >25/min, Altered mental awareness, Heart rate >120/min, Systolic blood pressure <100 mm Hg. iv) informed consent.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject enrolment will be based on adult patients presenting to the emergency department at the different sites with suspicion of organ dysfunction or identified at the hospital wars/units.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
infection-induced organ dysfunction | 72 hours
  To evaluate the presence or development of infection-induced organ dysfunction within a 72 hour time period from enrolment at the Emergency Department.

SECONDARY OUTCOMES:
To compare the specificity, sensitivity and accuracy of HBP against other biochemical markers | 72 hours
To investigate the specificity, sensitivity and accuracy in biochemical markers to predict mortality, ICU-care, days in hospital and the persistence of organ dysfunction. | 90 days
To investigate and identify risk factors for a negative long-term (5-10 year) outcome. | 10 years
• Organ dysfunction 24-36 and 72 hours after arriving at the hospital | 72 hrs
• Primary diagnosis infection (y/n) | 72 hrs
• number of days on ward and ICU | 90 days
• number of days of antibiotics , time to effective antibiotics | 72 hrs

CONTACTS AND LOCATIONS:
Locations (4):
- John Boyd, Vancouver, Canada
- Sweden (2):
  - Helsingborg, Helsingborg
  - Lund ED, Lund
- Bern ED, Bern, Switzerland